CLINICAL TRIAL: NCT07210086
Title: Phase II Non-Randomized Study Evaluating POSLUMA-PSMA PET Response After Oligo- Metastatic/Progressive-directed Treatment With Radiotherapy (PROMPT-R)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25339; P30CA033572 (NIH); NCI-2025-07236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25339 (Other: City of Hope Medical Center)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- De novo oligometastatic disease treated with ADT+ARSI+ablative intent RT (Other): De novo oligometastatic disease treated with ADT+ARSI+ablative intent RT and who have <=5 extrapelvic lesions detected on a baseline PSMA-PET and have rising PSA.
  Interventions: Drug: ADT; Drug: ARSI
- Recurrent disease with oligometastatic disease treated with ADT+ablative intent RT (Other): Recurrent disease with oligometastatic disease treated with ADT+ablative intent RT and who have <=5 extrapelvic lesions detected on a baseline PSMA-PET and have rising PSA.
  Interventions: Drug: ADT
- Recurrent prostate ca with oligometastatic disease who decline ADT/ARSI (Other): Recurrent prostate cancer with oligometastatic disease who decline ADT/ARSI and are treated with ablative intent RT alone and who have <=5 extrapelvic lesions detected on a baseline PSMA-PET and have rising PSA.
  Interventions: Other: No ADT/ARSI -decline

INTERVENTIONS:
Drug: ADT — Androgen Deprivation Therapy
  Arms: De novo oligometastatic disease treated with ADT+ARSI+ablative intent RT; Recurrent disease with oligometastatic disease treated with ADT+ablative intent RT
Drug: ARSI — Androgen Receptor Signaling Inhibitor
  Arms: De novo oligometastatic disease treated with ADT+ARSI+ablative intent RT
Other: No ADT/ARSI -decline — Recurrent prostate cancer with oligometastatic disease who decline ADT/ARSI and are treated with ablative intent RT alone and who have <=5 extrapelvic lesions detected on a baseline PSMA-PET and have rising PSA.
  Arms: Recurrent prostate ca with oligometastatic disease who decline ADT/ARSI

SUMMARY:
This study aims to evaluate the role of PSMA-PET and circulating tumor DNA (ctDNA) in monitoring prostate cancer progression and response to radiotherapy (RT). Specifically, it investigates how often early progression is detected on PSMA-PET before PSA rise, examines PET responses of lesions treated with RT at 6 and 12 months and their correlation with PSA changes and later progression, examines ctDNA changes following ablative-intent RT to metastatic sites, and explores the relationship between PSMA-PET radiological findings and ctDNA dynamics.

DETAILED DESCRIPTION:
Primary Objective:

* Identify the frequency of early progressive disease on PSMA-PET prior to PSA progression.

Secondary Objectives:

* Describe the PET response to lesions given RT at 6 months (and 12 month if applicable), and its relationship to PSA changes, and to later progressive disease both on PET and with PSA progression for each cohort
* Characterize the changes in ctDNA levels after ablative-intent RT to metastatic sites.
* Describe the radiological changes from PSMA-PET and its relationship with ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant or legally authorized representative.
* Age: ≥ 18 years
* KPS ≥ 70 or ECOG 0-1 (Appendix A)
* Biopsy-confirmed diagnosis of castration-sensitive prostate adenocarcinoma, as defined by rising PSA in setting of T>100
* Clinical diagnosis of de novo oligometastatic or oligoprogressive disease, as defined by one the following:

De novo oligometastatic: newly diagnosed prostate cancer AND ≤ five metastatic sites outside of the pelvis (Metastatic sites may not be brain or liver.) OR Hormone Sensitive Oligoprogressive: history of prior local therapy for prostate cancer AND ≤ five progressing metastatic sites outside of the pelvis (Metastatic sites may not be brain or liver.) AND Hormone sensitive defined as clinical progression in absence of castration (T>100)

* Measurable disease by PERCIST v1.0
* Eligible to receive ablative-intent radiation therapy (biologically effective dose [BED] >100, α/β ratio:2) directed to all sites of metastatic disease.
* Primary site of disease (Prostate +/- Seminal Vesicles) is controlled or will receive ablative intent treatment as a part of this treatment course.
* Baseline flotufolastat F18 PET imaging, if obtained as part of standard of care, is acceptable provided it was performed prior to the initiation of radiation therapy.
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 30 days after the last dose of protocol therapy. * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion CriteriPrior and concomitant therapies

* Any patient planning to receive lifelong continuous or intermittent ADT
* For the current treatment course, patient must not have received more than 3 months of neoadjuvant ADT prior to consent.
* Any contraindication to receiving flotufolastat F 18.
* Diagnosis of polymetastatic (newly diagnosed prostate cancer and more than five metastatic sites outside of the pelvis or metastatic sites in brain or liver.)
* Diagnosis of polyprogressive disease (History of metastatic prostate cancer with more than five progressive metastatic sites outside of the pelvis or metastatic sites in brain or liver).
* Patients with a history or evidence of HIV infection (unless on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial).
* Patients with history or evidence of chronic hepatitis B virus (HBV) infection (unless HBV viral load is undetectable on suppressive therapy).
* Patients with a history or evidence of hepatitis C virus (HCV) infection (unless treated and cured. Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Any contraindications to undergo PSMA-PET.
* Clinically significant uncontrolled illness.
* Other active malignancy. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2028-05-13 (Estimated); Study Completion 2028-05-13 (Estimated)

PRIMARY OUTCOMES:
Early PD on PSMA-PET prior to PSA-progression | Up to 5 years
  Estimate percentage of patients whose PSMA_PET shows progressing disease (either on new sites or previously irradiated sites) prior to PSA progression

SECONDARY OUTCOMES:
Describe the PET response to lesions and its relationship to PSA changes | Up to 5 years.
  Describe the PET response to lesions given RT at 6 months (and 12 months if applicable), and its relationship to PSA changes, and to later PD both on PET and with PSA progression for each cohort.
Characterize the changes in ctDNA levels | Up to 5 years.
  Characterize the changes in ctDNA levels after ablative-intent RT to metastatic sites and its relationship to PSMA-PET changes.

CONTACTS AND LOCATIONS:
Overall Officials: Rose Li, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Undecided